CLINICAL TRIAL: NCT02345408
Title: An Open-label Phase 1b Study to Evaluate the Safety and Efficacy of CCX872-B in Patients With Pancreatic Adenocarcinoma
Brief Title: Phase 1b Study of CCX872-B in Patients With Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL002_872
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCX872-B (Experimental): 150 mg once or twice daily given orally for at least 12 weeks
  Interventions: Drug: CCX872-B

INTERVENTIONS:
Drug: CCX872-B — Tablets (oral administration)

SUMMARY:
This is an open-label phase 1-b study to evaluate the safety and efficacy of CCX872-B in patients with pancreatic adenocarcinoma also receiving FOLFIRINOX chemotherapy.

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-resectable pancreatic adenocarcinoma with or without metastases
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2
* Anticipated life expectancy ≥ 12 weeks
* Radiographically measurable disease acc. to RECIST 1.1
* Use of adequate contraception (as described in protocol)
* Ability to provide written informed consent and comply with study requirements

Exclusion Criteria:

* Received other cancer treatment or investigational drug within 4 weeks prior to screening
* Women who are pregnant or breastfeeding
* Had major surgery within 4 weeks of first dose of study drug
* Inadequate liver, renal or bone marrow function within 2 weeks of first dose
* Serious concurrent illness, altered medical status or any uncontrolled medical condition
* Any infection requiring antibiotic or anti-viral treatment within 4 weeks of screening
* Known active HIV, HBV or HCV infection
* Inability to swallow tablets
* History or presence of any medical condition or disease which, in the opinion of the investigator, may place the subject at unacceptable risk for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02; Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 24 weeks
subject incidence of Grade 3 or 4 adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (2):
  - St Louis, Missouri
  - Rochester, New York
- Netherlands (4):
  - Amsterdam
  - Nijmegen
  - Netherland, Rotterdam
  - Sittard